CLINICAL TRIAL: NCT02526355
Title: Development and Assessment of a Mobile Phone Based Intervention to Reduce Maternal Depression and Improve Child Health
Acronym: TechMother
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TechMotherCare001
Record Dates: First submitted 2014-11-15; First posted 2015-08-18 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Maternal Depression
Keywords: Maternal depression; Mobile phone based intervention; Learning Through Play; CBT; Intelligent Real Time Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobile based Intervention (Experimental): Mobile based Intervention (Learning Through Play Plus) comprised of both LTP and CBT
  Interventions: Behavioral: Mobile based intervention
- Waiting List Control (No Intervention): Waiting List Control group will receive no intervention, but intervention will be offered to interested participants at the end of the study

INTERVENTIONS:
Behavioral: Mobile based intervention — Learning through Play Plus Intervention delivered through mobile phone
  Other Names: Intelligent Real Time Therapy iRTT
  Arms: Mobile based Intervention

SUMMARY:
The prevalence rate of maternal depression in Pakistani women and its effect on the growth and development of young children and child mortality is very high.

The main objective of this study is to increase access to evidence based psychological interventions for mothers who have children of age 0 to 30 months, consistent with her values. The study will be a 2 (conditions) into 3 (Time) single blind randomized controlled trail. Depressed mothers will be randomized either to intervention arm or control arm. Intervention will include text messages based on Learning Through Play Plus (LTP plus CBT).

DETAILED DESCRIPTION:
Disturbances in mother-infant relationship in depressed mothers negatively influence the child's development. There are a number of efficient treatments for postnatal depression including antidepressant medication, psychotherapy and psychosocial interventions. Tele-health and mobile health is a novel and emerging field in psychiatric and psychological care and treatment of mental health difficulties, it involves the use of telecommunications to provide health care, support and intervention from a distance.

The proposed study will test the efficacy of an innovative, affordable mobile based intervention program that can help mothers with postnatal depression in low resource countries such as Pakistan.

Participants will be recruited from maternal and child care centres in Karachi, Pakistan and those participants (n = 204) meeting inclusion criteria of the study will be randomized into one of the 2 treatment arms, i.e., intervention or control, after completion of baseline assessment. Intervention will be comprised of LTP Plus and will be delivered through text messages. Momentary Sampling assessment and Momentary Psychological intervention will be part of this study. Participants will be assessed again after completion of intervention (i.e., after 12 weeks) and then 3 months post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with mild to moderate depression will be included
* Mother of children age 0-30months
* The age range in the study is 18 to 44 years
* Participants having mobile phones will be included

Exclusion Criteria:

* Subjects will not be included if they had a diagnosed medical condition or significant physical or learning disability
* Any form of psychosis, or are currently under psychiatric care.
* Mothers with severe depression or suicidal ideation will not be included
* Mothers who will be receiving any psychological intervention will be excluded
* Mothers of children with any serious medical or psychiatric illness will also be excluded.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 208 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) | change in scores from baseline to 3rd month and 6th month
  EPDS will be used to screen depression in mothers with child 0-30 months.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | change in scores from baseline to 3rd month and 6th month
  PHQ-9 will be used to assess the severity of depression
EuroQoL-5 Dimensions (EQ-5D) | change in scores from baseline to 3rd month and 6th month
  EQ-5D will be used to assess the health related quality of life
Generalized Anxiety Disorder - 7 (GAD-7) | change in scores from baseline to 3rd month and 6th month
  GAD 7 will be used to assess severity of anxiety.
Knowledge of Expectation and Child Development | change in scores from baseline to 3rd month and 6th month
  25-item questionnaire will be used to assess maternal knowledge and expectations for child development in the first three years. Higher scores indicate better outcomes.
Clinical Interview Schedule Revised (CISR) | Change in scores from baseline to 3rd month and 6th month
  The clinical Interview Schedule-Revised is a structured diagnostic instrument that was developed from the Clinical Interview Schedule (CIS), to assess psychiatric problems
Assessment of the growth and development of children (Weight) | Change in scores from Baseline and 6 month
  Anthropometric measures of child growth will be collected through measuring children's weight in kilograms. weight and height will be combined to report BMI in kg/m^2
Assessment of the growth and development of children (Height) | Change in scores from Baseline and 6 month
  Anthropometric measures of child growth will be collected through measuring children height in meters. weight and height will be combined to report BMI in kg/m^2

OTHER OUTCOMES:
Client Satisfaction Questionnaire (CSQ) | 3rd month
  To assess participants' level of satisfaction with the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nusrat Husain, MD, Principal Investigator — University of Manchester
Locations (3):
- Pakistan (3):
  - Jinnah Hospital, Lahore, Punjab Province
  - Chiniot Maternity Hospital, Karachi, Sindh
  - Sobhraj Maternity hospital, Karachi, Sindh